CLINICAL TRIAL: NCT03789604
Title: A Multi-Center, Randomized, Double-Blind, Phase III Study of Platinum-Containing Chemotherapy With or Without CS1001 in Stage IV Non-Small Cell Lung Cancer Subjects
Brief Title: A Study of CS1001 in Subjects With Stage IV Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS1001-302
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CS1001 monoclonal antibody (Experimental)
  Interventions: Biological: CS1001 monoclonal antibody
- CS1001 placebo (Placebo Comparator)
  Interventions: Biological: CS1001 placebo

INTERVENTIONS:
Biological: CS1001 monoclonal antibody — Participant will receive CS1001 monoclonal antibody 1200 mg by intravenous infusion every 3 weeks, for up to 24 months; Drug Carboplatin on Day 1 of each 21-day cycle; Drug Pemetrexed on Day 1 of each 21-day cycle; Drug Paclitaxel on Day 1 of each 21-day cycle
  Arms: CS1001 monoclonal antibody
Biological: CS1001 placebo — Participant will receive CS1001 placebo 1200 mg by intravenous infusion every 3 weeks, for up to 24 months; Drug Carboplatin on Day 1 of each 21-day cycle; Drug Pemetrexed on Day 1 of each 21-day cycle; Drug Paclitaxel on Day 1 of each 21-day cycle
  Arms: CS1001 placebo

SUMMARY:
This is a multi-center, randomized, double-blind, phase III study to evaluate the efficacy and safety of CS1001 in combination with platinum-containing chemotherapy versus placebo in combination with chemotherapy in first-line treatment-naive subjects with stage IV non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in this trial; fully understand and informed of this trial, and able to provide written informed consent form (ICF).
2. 18-75 years of age (18 and 75 included) on the day of signing ICF.
3. Histologically or cytologically confirmed stage IV non-small cell lung cancer (staged according to the 8th International Association for the Study of Lung Cancer (IASLC) classification.
4. Subjects haven't received systemic treatment for advanced/metastatic NSCLC.
5. Measurable target lesion evaluated by investigators according to RECIST v1.1.
6. ECOG PS of 0-1.
7. Life expectancy ≥ 12 weeks.
8. Subject with prior anti-cancer treatment can only be enrolled when all toxicities except for hearing loss, alopecia and fatigue, of prior anti-cancer treatment has recovered to ≤ Grade 1 according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events (CTCAE) v4.03.
9. Subjects must have adequate organ function.
10. Women of childbearing potential (WOBPC, as defined in section 13.5) must have a negative pregnancy test ≤7 days prior to the first dose of investigational product. WOBCP or fertile men and their WOBCP partners must agree to use an effective method of birth control from providing signed ICF and for 6 months after last dose of investigational product.

Exclusion Criteria:

1. Histologically confirmed small cell lung cancer or containing small cell component.
2. Subjects with current active autoimmune disease or prior history of autoimmune disease.
3. Malignancies other than NSCLC within 5 years prior to randomization.
4. Known history of human immunodefiency virus (HIV) infection and/or acquired immune deficiency syndrome.
5. Subject with active hepatitis B or hepatitis C.
6. Subjects with known history of alcoholism or drugs abuse.
7. Has a known hypersensitivity to any component of study treatment, for example pemetrexed, cisplatin, carboplatin or other platinum compounds.
8. Subjects with other conditions that in the investigator's opinion may influence subject's compliance or make subjects not suitable for participating in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in all subjects evaluated by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | up to approximately 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 7 years
  OS defined as the time from randomization to all-cause death.
PFS assessed by BICR | up to approximately 5 years
  PFS defined as the time from randomization to the first occurrence of disease progression or all-cause death (whichever occurs first), as determined by the BICR according to RECIST v1.1
PFS in subgroup of participants with PD-L1 Expression≥1%, as determined by the investigator | up to approximately 5 years
  PFS after randomization as determined by the investigator according to RECIST v1.1 in the subgroup of patients with PD-L1 expression ≥1% defined by the SP263 immunohistochemistry (IHC) assay.
Objective Response Rate (ORR) assessed by the investigator according to RECIST v1.1 | up to approximately 5 years
  ORR, defined as the proportion of patients with a complete response (CR) or partial response (PR) on two consecutive occasions >=4 weeks apart, as determined by the investigator according to RECIST v1.1.
Duration of response (DOR) assessed by the investigator according to RECIST v1.1 | up to approximately 5 years
  DOR defined as the time between the date of the earliest qualifying response and the date of progressive disease or all-cause death, whichever occurs first, as determined by the investigator according to RECIST v1.1.
Safety and tolerability of CS1001 or placebo in combination with platinum-based chemotherapy | up to approximately 5 years
Pharmacokinetics (PK) and immunogenecity of CS1001 | up to approximately 5 years
Efficacy of CS1001 monotherapy in subjects cross over to receive CS1001 who experienced progressive disease after assigned to the placebo group in the double-blind phase (CS1001 or placebo in combination with chemotherapy) | up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhou C, Wang Z, Sun M, Cao L, Ma Z, Wu R, Yu Y, Yao W, Sun S, Chen J, Zhuang W, Cui J, Chen X, Lu Y, Shen H, Hu C, Liu J, Liu Y, Wang M, Li X, Sun P, Shu Y, Zhou J, Li J, Gu K, Wang C, Zhao H, Zhang Y, Liu C, Yang H, Zhang X, Ma R, Li L, Liang L, Li M, Wang J, Wang Q, Wang B, Dai H, Shi Q, Yang J. Sugemalimab versus placebo, in combination with platinum-based chemotherapy, as first-line treatment of metastatic non-small-cell lung cancer (GEMSTONE-302): 4-year outcomes from a double-blind, randomised, phase 3 trial. Lancet Oncol. 2025 Jul;26(7):887-897. doi: 10.1016/S1470-2045(25)00198-6. Epub 2025 Jun 13. PMID 40523368
- [Derived] Zhou C, Wang Z, Sun M, Cao L, Ma Z, Wu R, Yu Y, Yao W, Sun S, Chen J, Zhuang W, Cui J, Chen X, Lu Y, Shen H, Hu C, Liu J, Liu Y, Wang M, Li X, Sun P, Shu Y, Zhou J, Li J, Gu K, Wang C, Zhao H, Zhang Y, Liu C, Wang J, Chen R, Qin M, Wang H, Yang J. Interim survival analysis of the randomized phase III GEMSTONE-302 trial: sugemalimab or placebo plus chemotherapy as first-line treatment for metastatic NSCLC. Nat Cancer. 2023 Jun;4(6):860-871. doi: 10.1038/s43018-023-00578-z. Epub 2023 Jun 15. PMID 37322367
- [Derived] Zhou C, Wang Z, Sun Y, Cao L, Ma Z, Wu R, Yu Y, Yao W, Chang J, Chen J, Zhuang W, Cui J, Chen X, Lu Y, Shen H, Wang J, Li P, Qin M, Lu D, Yang J. Sugemalimab versus placebo, in combination with platinum-based chemotherapy, as first-line treatment of metastatic non-small-cell lung cancer (GEMSTONE-302): interim and final analyses of a double-blind, randomised, phase 3 clinical trial. Lancet Oncol. 2022 Feb;23(2):220-233. doi: 10.1016/S1470-2045(21)00650-1. Epub 2022 Jan 14. PMID 35038432